CLINICAL TRIAL: NCT00270426
Title: Benazepril for Advanced Chronic Renal Insufficiency
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Medical University, China (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SouthernMUC
Record Dates: First submitted 2005-12-23; First posted 2005-12-26 (Estimated); Last update posted 2006-05-05 (Estimated); Status verified 1999-03

CONDITIONS: Chronic Kidney Failure
Keywords: Advanced Chronic Renal Insufficiency; Benazepril
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — benazepril

INTERVENTIONS:
Drug: Benazepril

SUMMARY:
The purpose of this study is to further determine whether benazepril, could safely slow the progression of renal dysfunction in non-diabetic patients with advanced renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. serum creatinine concentration 1.5-5.0 mg/dL (133-442 µmol/L)
2. creatinine clearance 20 to70 mL/min/1.73 m2, with variations of less than 30 percent in the three months before the screening evaluation
3. non-diabetic renal disease
4. persistent proteinuria (defined as urinary protein excretion greater than 0.3 g/day for three or more months without evidence of urinary-tract infection or overt heart failure [New York Heart Association class III-IV]).

Exclusion Criteria:

* immediate need for dialysis; treatment with corticosteroids, non-steroidal anti-inflammatory drugs or immunosuppressive drugs; renovascular disease; myocardial infarction or cerebrovascular accident in the year preceding the trial; connective-tissue disease; obstructive uropathy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Fan Fan Hou, M.D.,Ph.D., Principal Investigator — Southern Medical University

REFERENCES:
- [Result] Hou FF, Zhang X, Zhang GH, Xie D, Chen PY, Zhang WR, Jiang JP, Liang M, Wang GB, Liu ZR, Geng RW. Efficacy and safety of benazepril for advanced chronic renal insufficiency. N Engl J Med. 2006 Jan 12;354(2):131-40. doi: 10.1056/NEJMoa053107. PMID 16407508
- [Derived] Vart P, Vaduganathan M, Jongs N, Remuzzi G, Wheeler DC, Hou FF, McCausland F, Chertow GM, Heerspink HJL. Estimated Lifetime Benefit of Combined RAAS and SGLT2 Inhibitor Therapy in Patients with Albuminuric CKD without Diabetes. Clin J Am Soc Nephrol. 2022 Dec;17(12):1754-1762. doi: 10.2215/CJN.08900722. Epub 2022 Nov 22. PMID 36414316